CLINICAL TRIAL: NCT01731327
Title: A Phase 1, Randomized, Open-Label, 2-Way Crossover Study To Evaluate The Pharmacokinetics (PK), Safety, And Bioavailability Of Tofacitinib Following Single Oral Dose Of MR 11 mg Compared To MR 22 mg In Healthy Volunteers
Brief Title: A Phase 1 Study To Evaluate The Pharmacokinetics (PK), Safety, And Bioavailability Of A Modified-Release (MR) Formulation Of Tofacitinib In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A3921132
Record Dates: First submitted 2012-11-14; First posted 2012-11-21 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: Phase 1; relative bioavailability; modified release; tofacitinib; CP-690; 550; pharmacokinetic
MeSH Terms: interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Treatment A (Experimental): A single dose of 11 mg tofacitinib modified-release (MR) administered in a fasting state.
  Interventions: Drug: tofacitinib modified-release (MR) formulation
- Experimental Treatment B (Experimental): A single dose of 22 mg tofacitinib modified-release (MR) administered in a fasting state.
  Interventions: Drug: tofacitinib modified-release (MR) formulation

INTERVENTIONS:
Drug: tofacitinib modified-release (MR) formulation — A single dose of 11 mg tofacitinib modified-release (MR) administered in a fasting state.
  Arms: Experimental Treatment A
Drug: tofacitinib modified-release (MR) formulation — A single dose of 22 mg tofacitinib modified-release (MR) administered in a fasting state.
  Arms: Experimental Treatment B

SUMMARY:
This study will explore the drug behavior and safety following single doses of tofacitinib modified-release (MR) 11 mg and MR 22 mg in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and/or healthy female subjects who are of non-childbearing potential.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease;
* Clinically significant infections within the past 3 months

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
AUCinf(dn): Area Under the Curve From Time Zero to Infinity, dose-normalized | 72 hours post dose
Cmax(dn): Maximum Observed Plasma Concentration (Cmax), dose normalized | 72 hours post dose

SECONDARY OUTCOMES:
AUClast(dn): Area Under the Curve From Time Zero to Last Quantifiable Concentration, dose normalized | 72 hours post dose
AUCinf: Area Under the Curve From Time Zero to Infinity | 72 hours post dose
Cmax: Maximum Observed Plasma Concentration | 72 hours post dose
AUClast: Area Under the Curve From Time Zero to Last Quantifiable Concentration | 72 hours post dose
Tmax: Amount of time drug takes to reach Cmax | 72 hours post dose
t ½: Terminal elimination half-life | 72 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921132&StudyName=A%20Phase%201%20Study%20To%20Evaluate%20The%20Pharmacokinetics%20%28PK%29%2C%20Safety%2C%20And%20Bioavailability%20Of%20A%20Modified-Release%20%28MR%29%20Formulation%20Of%20T